CLINICAL TRIAL: NCT00005276
Title: A Case Controlled Etiologic Study of Sarcoidosis (ACCESS)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1303
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2005-12

CONDITIONS: Lung Diseases; Sarcoidosis
MeSH Terms: conditions — Lung Diseases; Sarcoidosis

SUMMARY:
To test specific hypotheses concerning environmental, occupational, lifestyle, and other risk factors for sarcoidosis. Also, to examine the familial aggregation of sarcoidosis and to test genetic hypotheses concerning its etiology. Finally, to describe the natural history of sarcoidosis, particularly in African-Americans who appear to be disproportionately affected, and to implement a system for storing biological specimens including blood cells, plasma, and serum.

DETAILED DESCRIPTION:
BACKGROUND:

Sarcoidosis is a systemic granulomatous disorder of unknown etiology. While recognized as a distinct clinical entity for over a century, information on incidence, prevalence, risk factors, and natural history in the United States remains quite limited. Data available on the occurrence in the United States indicate that the incidence ranges from about 1 to 10 per 100,000 and prevalence from about 5 to 50 per 100,000. Incidence appears highest for young adults, ages 25 to 40, higher in females than males, and much greater in African Americans than other ethnic groups. Morbidity from this chronic disease is not well estimated by mortality data. In 1981, there were over 10,000 discharges from United States hospitals for sarcoidosis. Like mortality data, the hospital discharge information probably substantially underestimates the morbidity associated with sarcoidosis which is typically managed on an outpatient basis.

The Requests for Proposals were issued in September, 1994. Awards were made in June, 1995.

DESIGN NARRATIVE:

Each of ten clinical centers enrolled patients with sarcoidosis. Because population-based case-finding mechanisms have not been widely implemented for sarcoidosis, an institution-based rather than a population-based design was used. Participating institutions were located in geographic regions where the disease was known and ethnic and gender factors could be addressed. Several investigator-initiated studies were carried out.

In addition to etiology, ACCESS examined the socioeconomic status and clinical course of patients with sarcoidosis. Newly diagnosed cases of sarcoidosis were compared to age, sex, and race matched controls. Leads to the etiology of sarcoidosis have come from diverse sources: in clinical laboratory investigations, alveolitis has been found to precede granulomatous inflammation; in case control studies, familial aggregation has been identified; and in case reports, recurrence of granulomatous inflammation has been observed after lung transplantation.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-06; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baughman — University of Cincinnati; Michael Iannuzzi — Henry Ford Hospital; Marc Judson — Medical University of South Carolina; Genell Knatterud — Clinical Trials and Survey Corporation; Geoffrey McLennan — University of Iowa; David Moller — Johns Hopkins University; Lee Newman — National Jewish Center for Immunology & Respiratory Medicine; Milton Rossman — University of Pennsylvania; Alvin Teirstein — Icahn School of Medicine at Mount Sinai; Steven Weinberger — Beth Israel Hospital; Henry, Yeager — Georgetown University

REFERENCES:
- [Background] Gond NY, Khadabadi SS. Hepatoprotective Activity of Ficus carica Leaf Extract on Rifampicin-Induced Hepatic Damage in Rats. Indian J Pharm Sci. 2008 May-Jun;70(3):364-6. doi: 10.4103/0250-474X.43003. PMID 20046747
- [Background] Judson MA, Baughman RP, Teirstein AS, Terrin ML, Yeager H Jr. Defining organ involvement in sarcoidosis: the ACCESS proposed instrument. ACCESS Research Group. A Case Control Etiologic Study of Sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 1999 Mar;16(1):75-86. PMID 10207945
- [Background] Rybicki BA, Iannuzzi MC, Frederick MM, Thompson BW, Rossman MD, Bresnitz EA, Terrin ML, Moller DR, Barnard J, Baughman RP, DePalo L, Hunninghake G, Johns C, Judson MA, Knatterud GL, McLennan G, Newman LS, Rabin DL, Rose C, Teirstein AS, Weinberger SE, Yeager H, Cherniack R; ACCESS Research Group. Familial aggregation of sarcoidosis. A case-control etiologic study of sarcoidosis (ACCESS). Am J Respir Crit Care Med. 2001 Dec 1;164(11):2085-91. doi: 10.1164/ajrccm.164.11.2106001. PMID 11739139
- [Background] Baughman RP, Teirstein AS, Judson MA, Rossman MD, Yeager H Jr, Bresnitz EA, DePalo L, Hunninghake G, Iannuzzi MC, Johns CJ, McLennan G, Moller DR, Newman LS, Rabin DL, Rose C, Rybicki B, Weinberger SE, Terrin ML, Knatterud GL, Cherniak R; Case Control Etiologic Study of Sarcoidosis (ACCESS) research group. Clinical characteristics of patients in a case control study of sarcoidosis. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1885-9. doi: 10.1164/ajrccm.164.10.2104046. PMID 11734441
- [Background] Freemer M, King TE Jr. The ACCESS study: characterization of sarcoidosis in the United States. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1754-5. doi: 10.1164/ajrccm.164.10.2109111b. No abstract available. PMID 11734416
- [Background] Rossman M, Thompson B, Frederick M, Cizman B, Magira E, Monos D. Sarcoidosis: association with human leukocyte antigen class II amino acid epitopes and interaction with environmental exposures. Chest. 2002 Mar;121(3 Suppl):14S. doi: 10.1378/chest.121.3_suppl.14s. No abstract available. PMID 11893656
- [Background] Pandey JP, Frederick M; ACCESS Research Group. A Case Control Etiologic Study of Sarcoidosis. TNF-alpha, IL1-beta, and immunoglobulin (GM and KM) gene polymorphisms in sarcoidosis. Hum Immunol. 2002 Jun;63(6):485-91. doi: 10.1016/s0198-8859(02)00399-3. PMID 12039524
- [Background] Judson MA, Baughman RP, Thompson BW, Teirstein AS, Terrin ML, Rossman MD, Yeager H Jr, McLennan G, Bresnitz EA, DePalo L, Hunninghake G, Iannuzzi MC, Johns CJ, Moller DR, Newman LS, Rabin DL, Rose C, Rybicki BA, Weinberger SE, Knatterud GL, Cherniak R; ACCESS Research Group. Two year prognosis of sarcoidosis: the ACCESS experience. Sarcoidosis Vasc Diffuse Lung Dis. 2003 Oct;20(3):204-11. PMID 14620163
- [Background] Rossman MD, Thompson B, Frederick M, Maliarik M, Iannuzzi MC, Rybicki BA, Pandey JP, Newman LS, Magira E, Beznik-Cizman B, Monos D; ACCESS Group. HLA-DRB1*1101: a significant risk factor for sarcoidosis in blacks and whites. Am J Hum Genet. 2003 Oct;73(4):720-35. doi: 10.1086/378097. Epub 2003 Aug 20. PMID 14508706
- [Background] Newman LS, Rose CS, Bresnitz EA, Rossman MD, Barnard J, Frederick M, Terrin ML, Weinberger SE, Moller DR, McLennan G, Hunninghake G, DePalo L, Baughman RP, Iannuzzi MC, Judson MA, Knatterud GL, Thompson BW, Teirstein AS, Yeager H Jr, Johns CJ, Rabin DL, Rybicki BA, Cherniack R; ACCESS Research Group. A case control etiologic study of sarcoidosis: environmental and occupational risk factors. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1324-30. doi: 10.1164/rccm.200402-249OC. Epub 2004 Sep 3. PMID 15347561
- [Background] Taylor AN, Cullinan P. Sarcoidosis: in search of the cause. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1268-9. doi: 10.1164/rccm.2409006. No abstract available. PMID 15590884
- [Background] Rybicki BA, Walewski JL, Maliarik MJ, Kian H, Iannuzzi MC; ACCESS Research Group. The BTNL2 gene and sarcoidosis susceptibility in African Americans and Whites. Am J Hum Genet. 2005 Sep;77(3):491-9. doi: 10.1086/444435. Epub 2005 Jul 20. PMID 16080124
- [Background] Yeager H, Rossman MD, Baughman RP, Teirstein AS, Judson MA, Rabin DL, Iannuzzi MC, Rose C, Bresnitz EA, DePalo L, Hunninghakes G, Johns CJ, McLennan G, Moller DR, Newman LS, Rybicki B, Weinberger SE, Wilkins PC, Cherniack R; ACCESS Research Group. Pulmonary and psychosocial findings at enrollment in the ACCESS study. Sarcoidosis Vasc Diffuse Lung Dis. 2005 Jun;22(2):147-53. PMID 16053031
- [Background] Barnard J, Rose C, Newman L, Canner M, Martyny J, McCammon C, Bresnitz E, Rossman M, Thompson B, Rybicki B, Weinberger SE, Moller DR, McLennan G, Hunninghake G, DePalo L, Baughman RP, Iannuzzi MC, Judson MA, Knatterud GL, Teirstein AS, Yeager H Jr, Johns CJ, Rabin DL, Cherniack R; ACCESS Research Group. Job and industry classifications associated with sarcoidosis in A Case-Control Etiologic Study of Sarcoidosis (ACCESS). J Occup Environ Med. 2005 Mar;47(3):226-34. doi: 10.1097/01.jom.0000155711.88781.91. PMID 15761318
- [Background] Teirstein AS, Judson MA, Baughman RP, Rossman MD, Yeager H Jr, Moller DR; Case Control Etiologic Study of Sarcoidosis (ACCESS) Writing Group. The spectrum of biopsy sites for the diagnosis of sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 2005 Jun;22(2):139-46. PMID 16053030
- Available data/document: Individual Participant Data Set: ACCESS — http://biolincc.nhlbi.nih.gov/studies/access — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/access
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/access
- Available data/document: Procedures Manual — http://biolincc.nhlbi.nih.gov/studies/access